CLINICAL TRIAL: NCT01137253
Title: The Autonomic Nervous System, Nitric Oxide and TPA Interactions
Brief Title: Autonomic Nervous System and Nitric Oxide Interactions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Alfredo Gamboa, Research Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 091489
Record Dates: First submitted 2010-06-01; First posted 2010-06-04 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Endothelial Dysfunction
Keywords: Nitric Oxide; Autonomic Nervous System
MeSH Terms: interventions — Trimethaphan; Dental Occlusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trimethaphan (Experimental): Response to intrabrachial vasodilators during autonomic withdrawal
  Interventions: Drug: Trimethaphan
- Placebo (Placebo Comparator): Response to intrabrachial vasodilators during saline intravenous (IV) infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trimethaphan — Trimethaphan 4 mg/min IV, for the duration of the study (approximately 2 hours)
  Other Names: Blocked
  Arms: Trimethaphan
Drug: Placebo — Response to intrabrachial vasodilators during IV saline infusion
  Other Names: Intact
  Arms: Placebo

SUMMARY:
The investigators are interested in the role of the autonomic nervous system in the regulation of endothelial function among obese hypertensive subjects. In particular, the investigators will study how endothelial function (response to intra-arterial acetylcholine) changes during autonomic withdrawal.

ELIGIBILITY:
For lean healthy volunteers:

* 20 subjects (10 males and 10 females) aged 18-60 yr.
* All potential volunteers will have routine blood test to screen for hepatic, renal, and hematological abnormalities.
* Body mass index < 25Kg/m2 .
* Female volunteers of childbearing potential will undergo HCG pregnancy test at screening and again on the study day.

For Obese subjects with high blood pressure.

* 20 subjects (10 males and 10 females) aged 18-60 yr.
* All potential volunteers will have routine blood test to screen for hepatic, renal, and hematological abnormalities.
* Body mass index > 30 and less than 40 Kg/m2

  *High blood pressure (systolic=130 and diastolic = 85 mmHg)
* Female volunteers of childbearing potential will undergo serum HCG pregnancy test at screening and urine HCG pregnancy test again on the study day.

Exclusion criteria:

* Pregnant females
* Subjects unable to give voluntary informed consent
* Subjects on anticoagulant drugs or anemic
* Subjects with a recent medical illness
* Subjects with a history of coronary heart disease
* Subjects with known kidney or liver disease
* Subjects with recent weight loss or consuming low carbohydrate diet

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | 2 hours
  The dose response curve to intrabrachial vasodilators will be determined using the peak forearm blood flow during the last 5 minutes of each drug infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States